CLINICAL TRIAL: NCT03917121
Title: Pain Control of Needle-less Jet Anesthesia Versus Conventional Infiltration Anesthesia for Pulpotomy of Maxillary Primary Molars in Children: A Randomized Controlled Trial
Brief Title: Pain Control of Needle-free Versus Needle Injected Local Anesthesia for Pulpotomy of Upper Primary Molars in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lobna Salah El-Dien Mohamed Ahmed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2019-04-05
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Anesthesia, Local
Keywords: Jet anesthesia; Pressure anesthesia; Needle-free anesthesia; Needle-less anesthesia; Needle-free injection; Jet injection; Needle-less local anesthesia; Needle-less syringe; Needle infiltration anesthesia; Needle injection; Local infiltration anesthesia; Local anesthesia; Pulpotomy; Vital pulp therapy; Primary molars; Child patients; Pediatric patients; Children

STUDY DESIGN:
Intervention Model Description: Parallel group trial with a 1:1 allocation ratio
Who Masked: Outcomes Assessor
Masking Description: The duplicate outcome assessor (study director) and the assigned data analyst/ statistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Jet anesthesia (Experimental): Local infiltration anesthesia delivered using Madajet XL® (MADA Medical Products, Inc., Carlstadt, NJ, USA) needle-free jet injector
  Interventions: Device: Jet injector
- Conventional infiltration anesthesia (Active Comparator): Local infiltration anesthesia delivered using 25 gauged short needle attached, 1.8 ml carpule loaded standard metal dental syringe
  Interventions: Device: Needle attached dental syringe

INTERVENTIONS:
Device: Jet injector — * The injection site will be dried with a sterile cotton swab and benzocaine 20% topical anesthetic gel/ Opahl® (Dharma Research, Inc., Miami, FL, USA) will be applied to the site using a cotton applicator for 2 mins prior to injection.
  * Articaine hydrochloride 4% with epinephrine 1:100,000 anesthetic solution/ ARTINIBSA 4%® (Inibsa Dental S.L.U., Lliçà de Vall, Barcelona, Spain) will then be delivered using Madajet XL injector as per the manufacturer's instructions.
  * A classical formocresol pulpotomy treatment procedure will be performed using formocresol/ Pyrocresol® (Pyrax Polymars, Roorkee, Uttarakhand, India) for fixation and polymer reinforced zinc oxide-eugenol/ Zinconol® (PREVEST DentPro, Digiana, Jammu, India) for restoration.
  * Primary and secondary outcome variables will be measured and recorded via selected tools at pre-specified time points.
  * All treated molars will be finally restored with stainless steel crowns or definitive restorations as indicated.
  Other Names: Madajet XL needle-free injector; Needle-less syringe; Needle-less injector
  Arms: Jet anesthesia
Device: Needle attached dental syringe — * The injection site will be dried with a sterile cotton swab and benzocaine 20% topical anesthetic gel/ Opahl® (Dharma Research, Inc., Miami, FL, USA) will be applied to the site using a cotton applicator for 2 mins prior to injection.
  * Articaine hydrochloride 4% with epinephrine 1:100,000 anesthetic solution/ ARTINIBSA 4%® (Inibsa Dental S.L.U., Lliçà de Vall, Barcelona, Spain) will then be delivered using standard needle-attached syringe in a classical local infiltration.
  * A classical formocresol pulpotomy treatment procedure will be performed using formocresol/ Pyrocresol® (Pyrax Polymars, Roorkee, Uttarakhand, India) for fixation and polymer reinforced zinc oxide-eugenol/ Zinconol® (PREVEST DentPro, Digiana, Jammu, India) for restoration.
  * Primary and secondary outcome variables will be measured and recorded via selected tools at pre-specified time points.
  * All treated molars will be finally restored with stainless steel crowns or definitive restorations as indicated.
  Arms: Conventional infiltration anesthesia

SUMMARY:
This is a study that will be conducted on 6 to 8 years old children to compare the needle-less jet injector with the conventional needle attached syringe in terms of efficiency in controlling pain of local anesthetic infiltration and post-anesthetic pulpotomy of upper first primary molars. The study tests a null hypothesis that states that there is no difference in pain control efficiency of the compared anesthetic techniques when used for the selected treatment procedure in the specified population.

DETAILED DESCRIPTION:
* The conduct of this study is driven by the substantial advantages that are documented to be offered by jet anesthesia over needle injected anesthesia combined with the scarcity, heterogeneity, limitations and contradicting inconclusive results of previously conducted studies assessing the acceptance and anesthetic efficiency of jet injectors against conventional needle attached dental syringes in pediatric patients, particularly for pulpotomy of primary molars. Jet injection offers the opportunity to deliver local anesthesia without using a needle and hence helps to avoid all drawbacks associated with needle injection such as psychological distress; pain; inability to cope with dental treatment; prolonged chair-side time; avoidance of dental care; high clinician skills required for child management and needle-stick injuries. It also allows precise controlled dosing; fast delivery and onset of local anesthesia; absence of post-operative numbness and thus self-inflicted traumatic injuries; reduction of medical waste and cutting down of long-term costs on the clinician. However, the true adequacy of jet anesthesia necessary to complete dental treatment successfully and the acceptance of jet injection in a child patient is yet to be revealed through further research.
* This randomized controlled trial is to be performed on children attending the Diagnosis outpatient clinic in Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University, Egypt. Children will be screened via personal, medical and dental history taking from them and their parents/caregivers; clinical examination and radiographic examination to identify appropriateness for recruitment in the trial based on the pre-specified eligibility criteria. Legal guardians of eligible children will be informed of the trial aims, conditions and procedures in details and a written informed consent will be obtained from them upon agreement for their children to participate in the trial. A verbal assent will be also obtained from each potential participant following a simple explanation of the trial procedure.
* Based on the sample size to be calculated, a random allocation sequence will be computer generated and will be used to assign participants to the experimental group receiving jet anesthesia (group A) and the control group receiving conventional infiltration anesthesia (group B). The allocation sequence will be enclosed in sequentially numbered, opaque, sealed envelopes and disclosure of the randomization code to the principle investigator will be performed only upon allocation of each corresponding subject throughout the course of the trial.
* For each study group, participants will be introduced to the dental setting and dental instruments to be used and have the anesthetization and dental procedure simply explained while avoiding any anxiety-provoking words. Psychological behavior management techniques such as Tell-Show-Do, voice control, distraction and positive reinforcement will be used similarly for both study groups. Following delivery of anesthesia, pulpotomy of maxillary first primary molars will be performed.
* Throughout the treatment procedure, if rescue anesthesia was needed, it will be delivered by needle infiltration in both study groups and recorded.
* Primary and secondary outcome variables will be measured and recorded via selected tools at pre-specified time points.
* Definitive examination and diagnosis for determination of eligibility, anesthetization, treatment, outcome measurement and data collection procedures will be all performed by the principal investigator.
* The principal investigator will be responsible for managing any intervention-related harms encountered by participants, both medically and financially, following-up the participant whenever necessary and providing post-operative prevention and oral hygiene instructions.
* All examination charts and outcome sheets will be labelled each with a specific code unique to every individual participant. Participant personal information will be kept confidential in a secured limited access area. All data will be electronically backed-up and securely stored by the principal investigator. Statistical analysis and interpretation of the collected results will be performed.
* All study results are planned to be disclosed and communicated to the public via a written thesis that will be orally presented and discussed in a defense that is to be held in Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University, in the presence of a selected jury. A manuscript of the trial work is planned to be prepared and submitted for publication.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy (Classified as American Society of Anesthesiologists/ ASA I)
* Vital deeply carious maxillary first primary molars indicated for pulpotomy
* No previous dental experience
* Cooperative behavior (rating 3 or 4 on Frankl Category Rating Scale

Exclusion Criteria:

* Refuse to give assent to participate or have parents/caregivers refusing to sign the informed consent form

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Pain during pulpotomy score on Faces Pain Scale-Revised, aggregated by mean | Immediately following completion of pulpotomy procedure
  * Faces Pain Scale- Revised is a participant self-reported pain rating scale that consists of six line drawings of faces in different degrees of distress, scored along a 0-10 metric, measuring pain. The scale starts by a neutral face scored '0' representing no pain and ends with a frowning face scored '10' representing maximum pain. Scores increase in increments of 2.
  * The scale will be explained to the participant who will then be asked to choose the face that represents how much pain he/she feels. The pain score corresponding to the chosen face will be recorded.
Pain during pulpotomy score on Sound Eye Motor scale, aggregated by mean | Immediately following removal of dentin caries and initial access to pulp
  * Sound Eye Motor scale is a clinician-reported pain rating scale that considers three types of physical observations- sound, ocular and motor- and scores each along a 1-4 subscale, measuring pain.'1' is designated as comfort (represents no pain) and '4' is designated as painful (represents maximum pain). Scores increase in increments of 1.
  * The participant will be observed and a score will be given by the assessor on each of the three subscales. The three scores given will be summed to obtain the total pain score at a specific time point of interest.
  * Primary pain assessment on Sound Eye Motor scale will be performed by principal investigator and independent duplicate pain assessment on the same scale will be performed by study director.
Pain during pulpotomy score on Sound Eye Motor scale, aggregated by mean | Immediately following pulp extirpation
  * Sound Eye Motor scale is a clinician-reported pain rating scale that considers three types of physical observations- sound, ocular and motor- and scores each along a 1-4 subscale, measuring pain.'1' is designated as comfort (represents no pain) and '4' is designated as painful (represents maximum pain). Scores increase in increments of 1.
  * The participant will be observed and a score will be given by the assessor on each of the three subscales. The three scores given will be summed to obtain the total pain score at a specific time point of interest.
  * Primary pain assessment on Sound Eye Motor scale will be performed by principal investigator and independent duplicate pain assessment on the same scale will be performed by study director.

SECONDARY OUTCOMES:
Pain during injection score on Faces Pain Scale-Revised, aggregated by mean | Immediately following injection of local anesthesia
  * Faces Pain Scale- Revised is a participant self-reported pain rating scale that consists of six line drawings of faces in different degrees of distress, scored along a 0-10 metric, measuring pain. The scale starts by a neutral face scored '0' representing no pain and ends with a frowning face scored '10' representing maximum pain. Scores increase in increments of 2.
  * The scale will be explained to the participant who will then be asked to choose the face that represents how much pain he/she feels. The pain score corresponding to the chosen face will be recorded.
Pain during injection score on Sound Eye Motor scale, aggregated by mean | Immediately following injection of local anesthesia
  * Sound Eye Motor scale is a clinician-reported pain rating scale that considers three types of physical observations- sound, ocular and motor- and scores each along a 1-4 subscale, measuring pain.'1' is designated as comfort (represents no pain) and '4' is designated as painful (represents maximum pain). Scores increase in increments of 1.
  * The participant will be observed and a score will be given by the assessor on each of the three subscales. The three scores given will be summed to obtain the total pain score at a specific time point of interest.
  * Primary pain assessment on Sound Eye Motor scale will be performed by principal investigator and independent duplicate pain assessment on the same scale will be performed by study director.
Need for additional anesthesia, recorded as a binary (yes/no) outcome | Immediately following completion of treatment for participant
  Rescue anesthesia recorded by principal investigator

CONTACTS AND LOCATIONS:
Overall Officials: Lobna S. Mohamed, B.D.S., Principal Investigator — Cairo University; Randa Y. Abd Al Gawad, Ph.D., Study Chair — Cairo University; Mariam M. Aly, Ph.D., Study Director — Cairo University